CLINICAL TRIAL: NCT04368182
Title: A Study of AFP Specific T Cell Receptor Transduced T Cells Injection in Unresectable Hepatocellular Carcinoma
Brief Title: AFP Specific T Cell Receptor Transduced T Cells Injection(C-TCR055) in Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD7
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Autologous C-TCR055 administered by intravenous (IV) infusion
  Interventions: Biological: Autologous C-TCR055

INTERVENTIONS:
Biological: Autologous C-TCR055 — Autologous C-TCR055 administered by intravenous (IV) infusion

SUMMARY:
A study that aimed to assess the safety and anti-tumor activity of C-TCR055 injection in unresectable HCC patients

DETAILED DESCRIPTION:
This study plans to enroll 5 patients to assess the safety of C-TCR055. Subjects who meet the eligibility criteria will receive a single dose of C-TCR055 injection, and will be followed up post treatment for safety monitoring. The follow up period will last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to provide written informed consent. 2. Age 18-70 years old, male or female. 3. Patients must meet the following criteria:

  a. Histologically confirmed HCC; b. Serum AFP > 200ng/mL; c. Child-Pugh score ≤ 6; d. BCLC stage B and stage C defined by Chinese Liver Cancer Guideline 2017; e. Systemic therapy failed for HCC: those who received standardized systemic treatment for unresectable HCC and subsequently relapsed/progressed, or were intolerable or unwilling to receive treatment. Front-line system treatment should be approved in China (Sorafenib, lenvastinib, platinum-containing chemotherapy, regofinil); f. Previous systemic therapy was discontinued at least 2 weeks before apheresis; g. Local treatment (including surgery, ablation, interventional therapy, local radiotherapy, etc.) must be completed at least 4 weeks before apheresis, and there is no unhealed wound.

  4. Has at least 1 measurable lesion as defined per RECIST v1.1; 5. HLA-A 02:01 allele positive; 6. Liver AFP expression IHC tests
  1. ≥20% tumor cells positive, and ≤5% non-tumor tissue positive
  2. serum AFP ≥400ng/ml, and ≤5% non-tumor tissue positive. 7. ECOG score ≤ 1; 8. Expected survival > 12 weeks 9. Left ventricular ejection fraction (LVEF) ≥ 50% (measured by echocardiography). 10. No active pulmonary infections, normal pulmonary function and oxygen saturation ≥ 92% on room air 11. Laboratory criteria:

  <!-- -->

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  2. Platelets ≥ 60 x 10^9/L
  3. Hemoglobin ≥ 90g/L
  4. Serum total bilirubin ≤ 2 x ULN
  5. Aspartate aminotransferase (AST) and alanine aminotransferase
  6. Creatinine ≤ 1.5 x ULN 12.If patient has previous HBV infection, patient should receive antivirals treatment following treatment guidelines during study period, and the HBV DNA copies should below the detection limit at screening.

     13. Female subjects in childbearing age, their serum or urine pregnancy test must be negative, all subjects must agree to take effective contraceptive measures during the trial 14. Agree to abstain from alcohol during the study period 15. No contraindications for apheresis 16. Apheresis was received by laboratory, and passed QC.

     Exclusion Criteria:
* 1. Have a history of allergy to cellular products. 2. Subject has liver transplantation history. 3. tumor volume was greater than 70% of liver tissue 4. Main portal vein carcinoma thrombus 5. Medium to severe ascites 6. subjects received other anti-tumor systemic therapies which were not recommended in guidelines. Or subjects received immunocheckpoint inhibitors which were discontinued less than 6 weeks or 2 drug half-lives before apheresis.

  7. Subject has other primary cancer except for the following: A. Non-melanoma cured by excision, such as basal cell skin cancer. B.Cured in situ cancers such as cervical cancer, bladder cancer or breast cancer 8. Significant clinical gastrointestinal bleeding within 4 weeks before treatment. 9. Subjects with bone metastasis or central nervous system metastasis, or with hepatic encephalopathy, epilepsy, cerebrovascular accident and other central nervous system involvement diseases.

  10. Prior treatment with genetically modified T cell therapy or stem cell therapy.

  11. Uncontrolled active infection. Preventive antibiotics, antiviral and antifungal are permitted.

  12. Active hepatitis virus infection. HCV RNA positive. 13. Subjects with syphilis or other acquired, congenital immunodeficiency disorders, including, but not limited to, HIV infected persons, systemic lupus erythematosus, psoriasis, etc.

  14. Heart insufficiency subjects of Grade III or IV according to NYHA classification criteria.

  15. Subjects received systemic therapeutic steroid doses (except for the recent or current use of inhaled steroids) or other immunotherapy (such as interleukin-interferon, thymosin, etc.) within 2 weeks before Leukocyte apheresis 16. Subjects received radiotherapy within 6weeks before Leukocyte apheresis 17. Subjects who are pregnant, lactating, or pregnant within 6 months 18. Any other disease that may increase the risk of the subject or interfere with the results of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of C-TCR055 | start treatment to 12 months
  Determine if treatment with C-TCR055 is safe through assessment of adverse events(AEs) and serious adverse

SECONDARY OUTCOMES:
ORR | start treatment to 12 months
  Objective response rate based on RECIST v1.1
DCR | 3 months and 6 months
  Disease control rate based on RECIST v1.1
DOR | 12 months
  Duration of remission

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No